CLINICAL TRIAL: NCT05833841
Title: Assessment of Swallowing Function in Patients With Head and Neck Cancer Using Surface Electromyography and Video Fluoroscopy
Brief Title: Swallowing Function in Patients With Head and Neck Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HNQOL1
Record Dates: First submitted 2023-03-21; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Head Neck Cancer; Oral Cancer
Keywords: Swallowing; Aspiration; Surgery; treatment; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Deglutition Disorders | interventions — Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of swallowing function (Experimental): Measurement of swallowing function using Surface Electromyography and video flouroscopy
  Interventions: Diagnostic Test: Surface Electromyography and Video fluoroscopy

INTERVENTIONS:
Diagnostic Test: Surface Electromyography and Video fluoroscopy — Surface EMG of three muscle groups (masseter, submental, and infrahyoid) and video fluoroscopy with Omnipaque

SUMMARY:
Head and neck cancer (HNC) is the sixth most common cancer worldwide, accounting for 2.8% of all malignancies. The presence of tumor itself, as well as the treatment, can result in neuromuscular damage affecting any stage of the swallowing. Organ-sparing care has become more common in recent years, however, that this does not always imply functional preservation. Dysphagia and aspiration both can occur and can have complex causes. Normal swallowing has oral preparatory phase, pharyngeal phase, and the oesophageal phase, it is important to know what is the dysfunction and where. This study aim to evaluate the preoperative and postoperative swallowing function in patients with head neck cancer using electromyography (EMG) and video fluoroscopy.

DETAILED DESCRIPTION:
The process of swallowing includes the conscious effort to ingest food and a subconscious or reflex effort of bolus preparation. The preparation of the bolus is referred to as the preparatory phase, the transport of the bolus from the oral cavity and pharynx to the oesophagus as the transport phase and through the oesophagus as the oesophageal transport phase. The rhythm and pattern of the swallowing mechanism is controlled by a central pattern generator located in the medulla.

The tongue plays an important role in the preparatory phase by mixing the food and moving it towards the occlusal surface of the teeth. Sensory innervation across the oral mucosa and the tone of the facial muscles help in keeping the bolus within the oral cavity and in its manipulation. The soft palate approximates to the tongue to create a glossopalatal seal which prevents premature spillage in to the pharynx, while various movements of the mandible are imperative for the adequate grinding of the bolus. The tongue then contracts from anterior to posterior pushing the bolus back into the pharynx, the whole process taking about one second. This phase involves the Vth, VIIth and XIIth cranial nerves.

The pharyngeal phase is involuntary, with sensations travelling through the IXth and Xth cranial nerves and usually lasting one second. In this phase, the soft palate closes the nasopharynx, the larynx is elevated and closed, the pharyngeal constrictors contract and the cricopharynx relaxes. The true cords, the false cords, the epiglottis and the aryepiglottic folds constrict to form a barrier of several layers preventing aspiration.

The mechanism varies and there is no gold standard test that can accurately measure this dysfunction. Most patients are investigated only when it impairs the feeding and nasal feeding tubes are required. It is not know as to how much the function preserving conservative surgeries actually preserve the function and hence, the importance of this study.

ELIGIBILITY:
Inclusion Criteria:

* All Histologically proven cases of primary head and neck cancers.
* Head and neck cancer from stage T1 to T4a, N0 to N3, M0.
* Karnofsky performance status more than 70

Exclusion Criteria:

* Patients with neurological disease
* Pregnant and lactating women
* H/O any prior treatment such as Surgery, Chemotherapy, Radiotherapy Surgery for recurrent disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Swallowing dysfunction assessed by fluoroscopy and EMG | 6-8 weeks after surgery
  Aspiration is defined as leakage of dye in airway and dysphagia defined as difficulty in swallowing or hold up of contrast

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, Principal Investigator — Banaras Hindu University
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kronenberger MB, Meyers AD. Dysphagia following head and neck cancer surgery. Dysphagia. 1994 Fall;9(4):236-44. doi: 10.1007/BF00301917. PMID 7805423
- [Background] Dirix P, Nuyts S, Van den Bogaert W. Radiation-induced xerostomia in patients with head and neck cancer: a literature review. Cancer. 2006 Dec 1;107(11):2525-34. doi: 10.1002/cncr.22302. PMID 17078052
- [Background] Logemann JA, Rademaker AW, Pauloski BR, Lazarus CL, Mittal BB, Brockstein B, MacCracken E, Haraf DJ, Vokes EE, Newman LA, Liu D. Site of disease and treatment protocol as correlates of swallowing function in patients with head and neck cancer treated with chemoradiation. Head Neck. 2006 Jan;28(1):64-73. doi: 10.1002/hed.20299. PMID 16302193
- [Background] Al-Othman MO, Amdur RJ, Morris CG, Hinerman RW, Mendenhall WM. Does feeding tube placement predict for long-term swallowing disability after radiotherapy for head and neck cancer? Head Neck. 2003 Sep;25(9):741-7. doi: 10.1002/hed.10279. PMID 12953309
- [Background] Carrara-de Angelis E, Feher O, Barros AP, Nishimoto IN, Kowalski LP. Voice and swallowing in patients enrolled in a larynx preservation trial. Arch Otolaryngol Head Neck Surg. 2003 Jul;129(7):733-8. doi: 10.1001/archotol.129.7.733. PMID 12874074
- [Background] Kimata Y, Sakuraba M, Hishinuma S, Ebihara S, Hayashi R, Asakage T, Nakatsuka T, Harii K. Analysis of the relations between the shape of the reconstructed tongue and postoperative functions after subtotal or total glossectomy. Laryngoscope. 2003 May;113(5):905-9. doi: 10.1097/00005537-200305000-00024. PMID 12792331